CLINICAL TRIAL: NCT05689281
Title: T'Cher, Take Charge: Increasing PrEP Awareness, Uptake and Adherence Through Health Care Empowerment and Addressing Social Determinants of Health Among Racially Diverse Trans Women in the Deep South
Brief Title: Increasing PrEP With Trans Women in the Deep South
Acronym: T'Cher
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CrescentCare (Other)
Responsible Party: Principal Investigator, Narquis Barak, Principal Investigator, CrescentCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10275
Record Dates: First submitted 2023-01-06; First posted 2023-01-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be recruited on a rolling basis for a randomized, unblinded, cross-over stepped wedge study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP peer navigation (Experimental): Culturally informed health care empowerment and PrEP peer navigation and support through social determinant of health stressors
  Interventions: Behavioral: Peer PrEP Navigation

INTERVENTIONS:
Behavioral: Peer PrEP Navigation — Ecological momentary assessments to identify and address stressors related to social determinants of health (e.g., housing, substance use, mental health), and motivational interviewing to support participants' health care empowerment and progression along the PrEP continuum.

SUMMARY:
The goal of this to address barriers and facilitators to PrEP uptake, and encourage adherence among trans women via a single arm stepped wedge clinical trial. The main question is to compare PrEP uptake and adherence outcomes among trans women in the T'Cher intervention to the delayed study arm.

DETAILED DESCRIPTION:
The intervention will also assess changes in health care empowerment and support for Social Determinants of Health (SDoH) as mediating the effect of the intervention on PrEP uptake and adherence among trans women.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Declaration of willingness to comply with all study procedures and availability during the study
* Age 18 years old or older
* Male sex designated at birth
* Identify as trans woman, woman or another gender identity not associated with being a man
* Desire to use or re-start PrEP
* HIV uninfected
* Speaks English or Spanish
* Live in the New Orleans metropolitan statistical area (which includes 8 parishes)

Exclusion Criteria:

* Confirmed HIV infection by rapid algorithm testing and/or laboratory testing (described above)
* Prior or current participation in the active arm of an HIV vaccine trial with evidence of vaccine-induced seropositivity
* Concurrent or planned enrollment in a research study that provides PrEP
* Unwilling to attend quarterly follow-up visits, which will include survey participation
* Has any other condition which, based on the opinion of the investigator, would preclude provision of informed consent; make participation in the project unsafe; complicate interpretation of outcome data; or otherwise interfere with achieving the project objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans woman
Enrollment: 200 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | 24 months
  The proportion of participants enrolled in the study who begin to take PrEP
Social determinant stressors | 24 months
  The proportion of participants enrolled in the study who address social determinant stressors
Health care empowerment | 24 months
  The proportion of participants enrolled in the study who report improved healthcare empowerment

SECONDARY OUTCOMES:
Patterns and correlates of PrEP adherence | 24 months
  Analysis of PrEP adherence among those who begin PrEP. Patterns and correlates of adherence will be measures using data from self report surveys and urine assays

CONTACTS AND LOCATIONS:
Locations (1):
- NO/AIDS Task Force d.b.a. CrescentCare, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No